CLINICAL TRIAL: NCT05344703
Title: Is Y-Balance Test Predictive of Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Alex Habegger, Assistant Professor, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ArkansasCollegesHlthEd
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Concussion, Brain; Concussion; Eye
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Single group of 6th to 12th graders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Y Balance (Active Comparator): Subjects will perform Y-balance lower quarter
  Interventions: Diagnostic Test: Y balance
- Y Balance Plus Stroboscopic Glasses (Active Comparator): Subjects will perform Y-balance lower quarter with and without stroboscopic lenses
  Interventions: Device: Y Balance Plus Visual Perturbations

INTERVENTIONS:
Device: Y Balance Plus Visual Perturbations — Stroboscopic glasses will be added to the protocol for the participants to perform the Y-balance lower quarter to examine the differences in Y-balance scores as well as examining the Y-balance's ability to predict injury and concussion with visual perturbations.
  Arms: Y Balance Plus Stroboscopic Glasses
Diagnostic Test: Y balance — Subjects will perform Y-balance without any interventional strategies.
  Arms: Standard Y Balance

SUMMARY:
The Y Balance Test for the lower quarter (YBT-LQ) is a movement screen used to assess an athlete's risk for injury. The YBT-LQ is a dynamic balance test where the participant stands on a single leg and with the opposite lower extremity reaches are far in the anterior direction as they can, and this value is measured. The process is repeated in the posterior medial, and the posterior lateral directions. The final values are controlled for leg length of the participants. The YBT-LQ has been shown to be predictive of lower extremity injury in high school basketball players, but it is typically used as part of a battery of tests to determine the athlete's overall injury risk, but more questions remain to be answered. The research question: Is the YBT-LQ predictive of concussion in high school athletes? What are the norms for YBT-LQ in high school athletes? Does history of concussion effect YBT-LQ? Is the YBT-LQ with visual perturbations predictive of concussions? Is the YBT-LQ with visual perturbations predictive of lower extremity injury? What is the impact of visual perturbations on Y-balance and its injury prevention capability?

The target student participants will be 9th through 12th grade students; however, 6th to 8th grade students will be allowed to participate depending on the school or organization request. Informed consent will be obtained reiterating that participation is voluntary. Testing utilizing the YBT-LQ will occur, and sport of participation, age, height, weight, dorsiflexion, and leg length will be obtained. Follow up will be made via the athletic trainers and school personnel to indicate the effected athletes. Once the post-test follow up is complete athletes will be able to see their pre-test scores, and any questions will be answered at that time. This will be a longitudinal study where testing will take place at least two times per year, preferably three times per year over 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Participates in sport either school sanctioned or club

Exclusion Criteria:

* History of seizure

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-04 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Report of concussion in past year | 1 year
  Determine if patient sustained concussion since test date utilizing this questionnaire.
Report of lower extremity injury in past year | 1 year
  This will be determined utilizing intake questionnaire as developed by research team delineating joint or structure impacted by injury.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fort Smith Public Schools, Fort Smith, Arkansas
  - Greenwood Public Schools, Fort Smith, Arkansas

IPD SHARING:
Plan to Share IPD: No